CLINICAL TRIAL: NCT00674635
Title: A Randomized, Double-blind, Placebo-controlled, Bayesian Adaptive Dose Finding Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Repeat Intravenous Infusions GSK315234A in Patients With Active Rheumatoid Arthritis (RA)
Brief Title: Phase II Study Evaluating the Safety and Efficacy of GSK315234A in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 104972
Record Dates: First submitted 2008-04-22; First posted 2008-05-08 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: adaptive study,; DAS28,; monoclonal antibody; GSK315234A;; rheumatoid arthritis,
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo
- GSK315234A (Active Comparator): Part A single IV dose; Part B 3 repeat IV dose at Day 1, Day 28 and Day 56; Part C single SC dose
  Interventions: Drug: GSK3152314A

INTERVENTIONS:
Drug: GSK3152314A — Part A single IV dose; Part B 3 repeat IV dose at Day 1, Day 28 and Day 56; Part C single SC dose
  Arms: GSK315234A
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled adaptive, dose finding study to investigate the safety, tolerability, PK, PD and efficacy of single and repeat intravenous infusions of GSK315243A in patients with active rheumatoid arthritis. The study is divided into 2 parts: Part A is an adaptive, dose finding phase which will provide safety, tolerability, PK and PD on single intravenous infusions. Part B is a repeat dose phase which will provide safety, tolerability, PK, PD and efficacy following repeat intravenous infusions of a selected dose level.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 75 years of age, inclusive.
* All subjects must use acceptable contraception (as defined in the study restriction section) to ensure that no pregnancies occur during the course of the study and for at least 12 weeks after dosing for males and for 32 weeks after dosing for females (see Section 7.1 on contraception for more details).
* Body mass index within the range 18.5 - 35 kg/m2 inclusive, in addition to a weight range of 55 - 95kg.
* The subject must be capable of giving informed consent and can comply with the study requirements and timetable.
* The subject must have a diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology (ACR) (see Appendix 2).
* The subject must have a DAS28 disease activity score of greater than 4.2 at screening and pre-dose.
* The subject must have a CRP serum level of >/0.5mg/dl or an ESR level 28mm/hour at screening and pre-dose
* The subject has NOT received any biological therapy in the past, including biologicals for the treatment of rheumatoid arthritis
* The subject must have liver function tests including alanine transaminase (ALT) and aspartate transaminase (AST) within 1.5 times the upper limit of normal (ULN) and alkaline phosphatase (ALP) within 3 times ULN at screening. The patient must also have total bilirubin within the ULN at screening.
* The subject must have received at least 3 months of methotrexate and must be on a stable dose of methotrexate (up to 25 mg/week) for at least 8 weeks prior to screening and be willing to remain on this dose throughout the study.
* If sulfasalazine is being taken in addition to methotrexate, the subject must be on a stable dose for at least 4 weeks prior to screening and be willing to remain on this dose throughout the study.
* If hydroxychloroquine or chloroquine is being taken in addition to methotrexate, the subject must be on a stable dose for at least 3 months prior to screening and be willing to remain on this dose throughout the study.
* Those subjects on other oral anti-rheumatic therapies, which may include Non Steroidal Anti Inflammatory Drugs (NSAIDs), COX-2 inhibitors, oral glucocorticoids e.g. prednisolone (£10mg/day) must be on stable dosing regimens for at least 4 weeks prior to screening and be willing to remain on this regime throughout the study. Subjects receiving intramuscular glucocorticoids e.g methylprednisolone (£120 mg/month) must be on a stable dosing regimen for at least 3 months prior to screening and be willing to remain on this regimen throughout the study.
* The subject must be on a stable dose of folate supplements (5 mg/week) for at least 4 weeks prior to do

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination (e.g. haematology parameter outside the normal limits), or ECG (12 Lead or Holter).
* The subject has a positive Hepatitis B surface antigen or Hepatitis C antibody result at screening.
* The subject has a history of elevated liver function tests on more than one occasion (ALT, AST and ALP > 3 x Upper Limit of Normal (ULN); total bilirubin > 1.5 x ULN) in the past 6 months.
* Previous exposure or past infection caused by Mycobacterium tuberculosis
* The subject has an acute infection.
* The subject has a history of repeated, chronic or opportunistic infections that, in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as a participant in this trial.
* The subject has a history of malignancy, except for surgically cured basal cell carcinoma or females with cured cervical carcinoma (> 2 yrs prior).
* The subject has a history of human immunodeficiency virus (HIV) or other immunodeficiency disease.
* The subject whose calculated creatinine clearance is less than 50ml/min
* The subject has significant cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions that, in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as a participant in this trial.
* The subject has taken cyclosporine, leflonomide, cyclophosphamide or azathioprine within 1 month of screening. Subjects that have taken cyclosporine, leflonomide, cyclophosphamide or azathioprine in the past must have recovered from all drug related adverse events.
* The subject has taken gold salts or d-penicillamine within 1 month prior to screening. Subjects that have taken gold salts or d-penicillamine in the past must have recovered from all drug related adverse events.
* The subject has received intra-articular glucocorticoids within 1 month of screening.
* Recent history of bleeding disorders, anaemia, peptic ulcer disease, haematemesis or gastrointestinal bleeding
* Subjects with a history of haematological disease or acquired platelet disorders, including drug-induced thrombocytopaenia, acute idiopathic thrombocytopaenia or von Willebrand's disease.
* Subjects with a known risk of intra-cranial haemorrhage including Central Nervous System (CNS) surgery within the last 12 months, arterial vascular malformations, aneurysms, significant closed head trauma within 6 months or any other incident the investigator and/or medical monitor considers to be relevant.
* The subject has Hb <10 g/deciliter (dL) and platelet count < 150 x 109/Liter (L)
* Donation of blood in excess of 500 ml within a 56 day period prior to dosing
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the male subject to use a condom with spermicide in addition to having their female partner use another form of contraception such as an interuterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants of levonorgestrel or a tubal ligation if the woman could become pregnant for at least 12 weeks after dosing
* An unwillingness of female subject of child bearing potential to use adequate contraception, as defined in the study restriction section. If necessary, women of non-child bearing potential (i.e. post-menopausal or surgically sterile e.g. tubal ligation or hysterectomy or bilateral oophorectomy) will be confirmed. Postmenopausal status will be confirmed by serum follicle stimulating hormone (FSH) and oestradiol concentrations at screening. Surgical sterility will be defined as females who have had a documented hysterectomy, tubal ligation or bilateral oophorectomy.
* The subject has a history of use of drugs of abuse within 12 months prior to screening.
* History of regular alcohol consumption exceeding average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). Subjects who regularly consume more than 12 units of alcohol in a 24h period will also be excluded. 1 unit is equivalent to a half-pint (220ml) of beer/lager or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* Positive pregnancy test or lactating at screening.
* Participation in a trial with any investigational drug within 3 months or 5 half-lives (whichever is longer) before

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
• To assess the safety and tolerability of GSK315234A after single and repeat intravenous infusions in subjects with active rheumatoid arthritis on a background of methotrexate. | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
  safety assessment includes AEs, vital signs, ECG, clinical laboratory tests.
• To assess the effect of GSK315234A on disease activity [as defined by Disease Activity Score (DAS) 28 score] on Day 28 after a single intravenous infusion | Part A total of 150 days
  DAS28 at Day 28 and DAS28 at Day 56
• To assess the effect of GSK315234A on disease activity [as defined by Disease Activity Score (DAS) 28 score] on Day 56 in subjects with active rheumatoid arthritis on a background of methotrexate (Part B and Part C). | Part B total of 236 days and Part C total of 180 days
  DAS28 scores on Day 56 (Part B and C)

SECONDARY OUTCOMES:
Weighted mean DAS28 after single and repeat intravenous doses | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Plasma PK parameters of GSK315234A after single and repeat intravenous doses including free, and bound GSK315234A (serum) concentrations, AUC(0-¥), Cmax, clearance, volume of distribution and accumulation ratio | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
DAS28 and EULAR response criteria after single and repeat intravenous doses | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
ACR20/ACR50/ACR70 response after single and repeat intravenous doses | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Number of swollen joints assessed using 28-joint counts. | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Number of tender/painful joints assessed using 28-joint counts. | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Subject's pain assessment | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Physician's global assessment of arthritis condition. | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Patients' global assessment of arthritis condition. | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Functional disability index (Health Assessment Questionnaire) | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
C-reactive Protein (CRP). | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
ESR | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Global Fatigue Index | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
HAQ disability index | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Pharmacodynamic biomarkers after single and repeat intravenous doses: | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Characteristic AUC50 and EC50 for clinical endpoint changes with plasma exposure model, as assessed by sigmoid Emax and indirect response PK/PD models. | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
Immunogenicity (Human anti-GSK315234A antibodies) | Part A total of 150Days; Part B total of 236 days and Part C total of 180 days
• To assess the relative bioavailability of GSK315234A administered subcutaneously (Part C) as compared to intravenous administration in subjects with active rheumatoid arthritis on a background of methotrexate | Part C total of 180days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Australia (3):
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- New Zealand (3):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Wellington
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yaroslavl
- Serbia (2):
  - GSK Investigational Site, Belgrade
  - GSK Investigational Site, Niška Banja
- Ukraine (4):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Choy EH, Bendit M, McAleer D, Liu F, Feeney M, Brett S, Zamuner S, Campanile A, Toso J. Safety, tolerability, pharmacokinetics and pharmacodynamics of an anti- oncostatin M monoclonal antibody in rheumatoid arthritis: results from phase II randomized, placebo-controlled trials. Arthritis Res Ther. 2013 Sep 24;15(5):R132. doi: 10.1186/ar4312. PMID 24286335
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 104972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register